CLINICAL TRIAL: NCT00392717
Title: Effect of Atorvastatin and Fish Oils on Lipoprotein Metabolism in Visceral Obesity
Brief Title: Regulation of Lipoprotein Metabolism in Obese Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: EC-576
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Obesity; Dyslipidemia; Insulin Resistance
Keywords: lipoprotein metabolism; cardiovascular disease; obesity
MeSH Terms: conditions — Obesity; Dyslipidemias; Insulin Resistance; Cardiovascular Diseases | interventions — Atorvastatin; Fish Oils

INTERVENTIONS:
Drug: Atorvastatin
Drug: Fish oils

SUMMARY:
Visceral obesity is strongly associated with dyslipidaemia (hypertriglyceridaemia, low HDL-cholesterol and mildly elevated LDL-cholesterol) and insulin resistance, key characteristics of metabolic syndrome (MetS). Recent evidence has clearly established that the risk of CVD is increased in subjects with the MetS. The precise reason for this remains unclear, but appears to be closely related with dyslipidaemia. Effective management of dyslipidaemia is important to reduce the risk of CVD in these subjects.

Hypothesis: Inhibition of hepatic cholesterol synthesis by statins and triglyceride synthesis by fish oils improve lipoprotein metabolism in visceral obese men.

DETAILED DESCRIPTION:
The study employed a factorial study design, stable isotopy and mathematical modelling to examine the independent and combined effects of decreasing cholesterol substrate availability with atorvastatin and decreasing triglyceride substrate availability with fish oils on lipoprotien kinetics (apoB, apoA, apoC-III and chylomicron remnants) in insulin-resistant men with visceral obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obesity was defined as a waist circumference >100 cm, waist:hip ratio >0.97 and BMI >29 kg/m2.
* Subjects were selected for having insulin-resistance, defined as a homostasis model assessment (HOMA) score (21) >5.1 (i.e. one SD above the mean for a reference population of 22 lean, normolipidemic healthy males of similar age).
* All subjects had plasma triglyceride >1.2 mmol/L and cholesterol >5.2 mmol/L at screening while consuming ad libitum, weight-maintaining diets

Exclusion Criteria:

* diabetes mellitus, apolipoprotein E2/E2 genotype, macroproteinuria, creatinemia, hypothyrodism, or abnormal liver enzymes.
* Subjects did not consume fish oil supplements or drank more than 30g alcohol/day.
* None reported a history of CVD, or was taking medication or other agents known to affect lipid metabolism.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 1998-02; Study Completion 2002-03

PRIMARY OUTCOMES:
Fractional catabolic rate of apoB, apoA, apoC-III and chylomicron remnants (before and after 6 week treatments)
Production rate of apoB, apoA, apoC-III and chylomicron remnants (before and after 6 week treatments)

SECONDARY OUTCOMES:
Cholesterol
Triglyceride
LDL-cholesterol
Adipocytokines
Genetic polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Dick C Chan, PhD, Principal Investigator — The University of Western Australia; Gerald F Watts, MBBS PhD, Study Chair — The University of Western Australia; P Hugh H Barrett, PhD, Study Director — The University of Western Australia
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Chan DC, Barrett PH, Ooi EM, Ji J, Chan DT, Watts GF. Very low density lipoprotein metabolism and plasma adiponectin as predictors of high-density lipoprotein apolipoprotein A-I kinetics in obese and nonobese men. J Clin Endocrinol Metab. 2009 Mar;94(3):989-97. doi: 10.1210/jc.2008-1457. Epub 2008 Dec 30. PMID 19116237